CLINICAL TRIAL: NCT00882076
Title: Clofarabine, Etoposide, and Mitoxantrone for Relapsed and Refractory Acute Leukemias
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study closed prematurely
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, David F. Claxton, MD, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-096
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Leukemia
Keywords: acute lymphoblastic leukemia; chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Clofarabine; Mitoxantrone; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Treatment Cohort 1 (Experimental): Etoposide (Days 1-5) 100 mg/m2; Mitoxantrone (Days 1-3) 8 mg/m2 (3 doses); Clofarabine (Days 2-6) 20 mg/m2
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone; Drug: Etoposide
- Treatment Cohort 2 (Experimental): Etoposide (Days 1-5) 100 mg/m2; Mitoxantrone (Days 1-3) 8 mg/m2; Clofarabine (Days 2-6) 25 mg/m2
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone; Drug: Etoposide
- Treatment Cohort 3 (Experimental): Etoposide (Days 1-5) 100 mg/m2; Mitoxantrone (Days 1-3) 8 mg/m2; Clofarabine (Days 2-6) 30 mg/m2
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone; Drug: Etoposide
- Treatment Cohort 4 (Experimental): Etoposide (Days 1-5) 100 mg/m2; Mitoxantrone (Days 1-5) 8 mg/m2; Clofarabine (Days 2-6) 30 mg/m2
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone; Drug: Etoposide
- Treatment Cohort 0 (Experimental): Etoposide (Days 1-5) 100 mg/m2; Mitoxantrone (Days 1-3) 8 mg/m2; Clofarabine (Days 2-6) 10 mg/m2 (In the event of a DLT in Treatment Cohort 1)
  Interventions: Drug: Clofarabine; Drug: Mitoxantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Clofarabine — For Treatment Clofarabine will be administered on Days 2-6 at the dose of 20mg/m2 in Cohort 1, 25mg/m2 in Cohort 2 and 30mg/m2 in Cohort 3 and 4 and 10mg/m2 in Cohort 0 (In the event of excessive DLT in Treatment Cohort 1). For Retreatment Clofarabine will be administered on Days 1-4 at the dose of 20mg/m2 in Cohort 1, 25mg/m2 in Cohort 2 and 30mg/m2 in Cohort 3 and 4 and 10mg/m2 in Cohort 0 (In the event of excessive DLT in Retreatment Cohort 1).
  Other Names: Clolar
Drug: Mitoxantrone — For Treatment Mitoxantrone will be administered on Days 1-3 at the dose of 8mg/m2 in Cohort 1, 2, 3 and on Days 1-5 for Cohort 4 and on Days 1-3 8mg/m2 in Cohort 0 (In the event of excessive DLT in Treatment Cohort 1). For Retreatment Mitoxantrone will be administered on Days 1-2 (2 doses) at the dose of 8mg/m2 in Cohort 1, 2 and 3 and on Days 1-4 (4 doses) at the dose of 8mg/m2 in Cohort 4, and on Days 1-2 (2 doses) at the dose of 8mg/m2 in Cohort 0 (In the event of excessive DLT in Retreatment Cohort 1).
  Other Names: Mitoxantrone hydrochloride
Drug: Etoposide — For Treatment Etoposide will be administered on Days 1-5 at the dose of 100mg/m2 in Cohort 1, 2, 3, 4 and Cohort 0 (in the event of excessive DLT in Treatment Cohort 1). For Retreatment Etoposide will be administered on Days 1-4 at the dose of 100mg/m2 in Cohort 1, 2, 3, 4 and Cohort 0 (in the event of excessive DLT in Retreatment Cohort 1).
  Other Names: Etoposide Phosphate

SUMMARY:
The purpose of this study is to establish toxicity and a maximum tolerated dose recommended phase 2 dose of Clofarabine in combination with Etoposide and Mitoxantrone for therapy of relapsed or refractory acute leukemias. The investigators will observe responses with these therapy agents and assess the impact of Clofarabine interacting with Etoposide in induction of DNA strand breaks.

DETAILED DESCRIPTION:
This will be a phase I study with a standard 3x3 design. Patients will proceed to treatment through a series of cohorts with the three drugs being delivered over five days beginning with a dose of Etoposide 100 mg/m2 on days 1-5,Mitoxantrone 8 mg/m2 days 1-3, and clofarabine at 20 mg/m2 IV on days 2-6. Presuming this and subsequent cohorts are tolerable and no more than 1 patient per cohort develops DLT, MTD patients will be treated in cohorts of 3-6 patients up to a final dose level of Etoposide 100 mg/m2 on days 1-5,Mitoxantrone 8 mg/m2 days 1-5, and Clofarabine at 30 mg/m2 IV on days 2-6. Patients failing to enter remission may receive 4 days of therapy with Etoposide 100 mg/m2 on days 1-4,Mitoxantrone 8 mg/m2 days 1-2 or 1-4,and Clofarabine at 20-30 mg/m2 IV on days 1-4. According to established definitions for dose limiting toxicity a recommended phase II dose will be established. After this is established the final cohort will be expanded to 15 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adequate renal and hepatic function.
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
* LVEF must be ≥ 50% within 2 weeks.

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up or interpretation of study results.
* Have had a diagnosis of another malignancy, unless the patient has been disease free for at least 3 years following the completion of curative intent therapy with the following exceptions: patients with treated non-melanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for the study if definitive treatment for the condition has been completed. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed. Additionally, patients with prostate cancer treated with radiation therapy are also eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Establish toxicity of Clofarabine in combination with Etoposide and Mitoxantrone for therapy of relapsed or refractory acute leukemias | Days 30-45
Establish dose limiting toxicity of Clofarabine in combination with Etoposide and Mitoxantrone for therapy of relapsed or refractory acute leukemias | Days 30-45
Establish maximum tolerated dose recommend Phase 2 dose of Clofarabine in combination with Etoposide and Mitoxantrone for therapy of relapsed or refractory acute leukemias | Days 30-45

SECONDARY OUTCOMES:
Observe response of relapsed or refractory acute leukemias to therapy with these agents. | 30-70 days
Assess the impact of Clofarabine interacting with Etoposide and Mitoxantrone in induction of DNA strand breaks | 30-45 days

CONTACTS AND LOCATIONS:
Overall Officials: David F. Claxton, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Determine if data is valuable